



# PARTICIPANT INFORMATION SHEET & CONSENT FORM

NUS-IRB Reference Code: NUS-IRB-2023-859

#### 1. Protocol title

Exploring the Role of Parental Emotion Regulation and Outcomes of Parental Emotional Coaching on Child and Adolescent Psychosocial Outcomes

# 2. Principal Investigator and co-investigator(s), if any, with the contact number and organization:

Principal Investigator: Ong Jiehan Jamie Organization: National University of Singapore

Email: psyoj@nus.edu.sg

Co-Investigator: Dr Ryan Y. Hong

Organization: National University of Singapore Phone: 65166120; Email: <a href="mailto:ryan.hong@nus.edu.sg">ryan.hong@nus.edu.sg</a>

Co-Investigator: Dr Chee Tji Tjian

Organization: National University Hospital Systems

Email: tji tjian chee@nuhs.edu.sg

Co-Investigator: Dr Tan Poh Lin

Organization: National University Hospital Systems

Email: poh lin tan@nus.edu.sg

Co-Investigator: Dr Chin Zhen Hui (PsyD)

Organization: National University Hospital Systems

Email: zhen hui chin@nuhs.edu.sg

Co-Investigator: Ng Min Geng

Organization: National University of Singapore

Email: mingeng@u.nus.edu

## 3. What is the purpose of this research?

You are invited to participate in a research study. This information sheet provides you with information about the research study. The Principal Investigator (the person in charge of this research) or his/her representative will also describe this research to you and answer all of your questions. Read the information below and ask questions about anything you don't understand before deciding whether to take part.

The purpose of this research is to examine how parental emotional regulation and emotion coaching strategies affect children's psychosocial outcomes. This research is conducted in partial fulfilment of the requirements of the Principal Investigator's Ph.D. (Psychology) degree.

# 4. Who can participate in the research? What is the expected duration of my participation? What is the duration of this research?

To be eligible for this research, the child in the family must be between 7 to 17 years old. One parent and one child are required to take part in the research together. Only one





child per family is allowed for participation. Parents and children need to be proficient in English. Children and parents with physical impairments (apart from corrected vision), psychotic symptoms, known neurodevelopmental disorders or severe mood disorders, are not eligible.

This study has 2 parts. If you are only interested in Study 1, you will only be required to respond to a set of questionnaires at Timepoint 1. If you are interested in Study 2, it will span across 9 to 10 weeks, with parents and children responding to survey at 3 timepoints, which as roughly 1 month apart. They will be informed to complete the questionnaire at 3 specific time points, i.e. at beginning of study is Timepoint 1 (T1), 1-month after T1 and 2-month after T1. Each time it will take approximately 30 minutes (for parent) and 15 minutes (for child) to complete the questionnaire.

In Study 2, the parent will be invited to join a 3-hour parent workshop once. After which, they will be offered 2 individual Zoom/phone consultations with a psychologist.

The duration of the entire research study is 2 years.

5. What is the approximate number of research participants involved? We aim to recruit 400 participants (or 200 parent-child dyads).

## 6. What will be done if I take part in this research study?

This study has 2 parts. If you take part in Study 1, you and your family (i.e., 1 parent and 1 child) will only need to complete 1 set of questionnaires. It will take 30 minutes (for parent) and 15 minutes (for child) to complete the questionnaire. You are required to complete the questionnaire sets in one sitting. You are encouraged to take breaks when needed. There is no limit to the number of breaks that you may take. Parent and child can complete the questionnaires at their own time, it does not have to be completed concurrently.

Participants' responses on the respective questionnaire sets would be kept strictly confidential and not revealed to other members of their family. If the child requires assistance to complete the questionnaire, the parent may assist or reach out to the researcher for assistance. Participants are encouraged to not skip any questions and a copy of the questionnaire will be shown to you before consent is given.

Here are some examples of the questions:

- "I find it hard to wind down."
- "Mv child thinks about/I think about death."
- "I felt that life was meaningless."
- "The responsibility of being a parent seems like too much for me."

If you have indicated interest to participate in Study 2, parents will attend a 3-hour parent workshop as part of the study. For this part of the study, parents will be randomly assigned into 2 groups – 1. Emotion Coaching Group and 2. Waitlist Control Group. You will not know which group you will be assigned to. Parent and child will then have to complete a set of questionnaires at another 2 timepoints. After you have completed the study, the researcher will provide a debrief.

Some research designs require that the full extent of the study not be explained prior to participation. Although we have described the general nature of the tasks that you will be asked to perform, the full intent of the study will not be explained to you until after the completion of the study. At that time, we will provide you with a full debriefing which will include an explanation of the hypothesis that was tested and other relevant background information pertaining to the study. You will also be given an opportunity to ask any questions you have about the hypothesis and the procedures used in the study.





# 7. How will my privacy and the confidentiality of my research records be protected?

Only the principal investigator, co-investigators, and research assistants in this study will have access to your personal data (e.g. names and contact information) for the purpose of contacting you to provide information regarding the study. Personal data will never be used in a publication or presentation.

Personal data collected refers only to the parents/guardians as the children's data will be tagged to theirs, so that no personal data (other than names) will be collected from the minors, and all contacting will be done via their parents.

All identifiable research data will be coded (i.e. only identified with a code number) at the earliest possible stage of the research. The coded data may be shared with the funding organisation upon their requests. The code key will be held by the PI.

Personal data will be discarded once the data are fully analysed and will not be used for future research. Your participation does not involve information in individually identifiable form. The code key will also be discarded together with the personal data.

All data collected will be kept in accordance with the University's Research Data Management Policy. Research data used in any publication will be kept for a minimum of 10 years before being discarded.

## 8. What are the possible discomforts and risks for participants?

During the parent workshop, parents might get emotional when sharing about their difficulties. The workshop facilitators are either trained psychologists or psychologist trainees, and all are/will be equipped to manage such situations. Probability and magnitude of this risk is low.

Minors may feel pressured to answer the questionnaires in specific ways in the presence of their parents, they will be informed of the above confidentiality procedures and be allowed to skip questions they are uncomfortable with.

If scores on the questionnaires reflect concerning behaviors or mental health issues in both parent and child, the researchers, who are trained psychologists or psychologist trainees, will reach out to the parents to determine continuation of the research and whether a direct referral to relevant professional services may be required.

Similarly, if during the workshop, the trained professionals determine that the parents/child may need longer term intervention, they will be directed to relevant external professional services. A list of these services and resources will be provided to you (and to keep) at the end of each completed guestionnaire.

No other physical or psychological discomfort is known to be associated with this study.

#### 9. What is the compensation for any injury?

No injury and/or compensation are expected for participation in this study.

# 10. Will there be reimbursement for participation?

You and your family will be reimbursed up to SGD60 for your participation. Specifically, each member of the family will be reimbursed SGD10 per wave for completion of his/her respective questionnaire set. Do note that each individual will have to complete all the compulsory questions in his/her respective questionnaire set in order for him/her to receive the reimbursement. Participants who only agree to participate in Study 1, will only receive reimbursement for questionnaires completed at the beginning of the study.





For the entire study (Study 1 and 2), there will be 3 waves of questionnaires administered, 3 questionnaires per wave (1 for the child and 1 for the parent).

Please refer to table below for an example of the reimbursement schedule. Note that the timing for the administration of the questionnaires are an approximate.

| Estimated Timepoints | Parent | Child |
|----------------------------|-------------------|-------------------|
| At the beginning of the | Questionnaire 1 – | Questionnaire 1 – |
| study | Reimbursed SGD10 | Reimbursed SGD10 |
| 1 month after the parent | Questionnaire 2 – | Questionnaire 2 – |
| workshop OR 1 month | Reimbursed SGD10 | Reimbursed SGD10 |
| later | | |
| 1-month after completing | Questionnaire 3 – | Questionnaire 3 – |
| the 2 <sup>nd</sup> set of | Reimbursed SGD10 | Reimbursed SGD10 |
| questionnaires | | |

# 11. What are the possible benefits to me and to others?

The knowledge gained from this study may provide valuable directions in tailoring familiar and parental support available in the community and clinical setting. It could also provide a stepping stone to further develop research and services in the area of children and adolescent with emotional and behaviour difficulties.

In addition, complimentary parent workshops and brief psychological consultations will be provided, to equip parents with various strategies to manage their children's emotions and behaviours. There are no direct benefits to participants who did not participate in the parent workshops.

### 12. Can I refuse to participate in this research?

Yes, you can. Your decision to participate in this research study is voluntary and completely up to you and your family. You and your family can also withdraw from the research at any time without giving any reasons, by informing the principal investigator and all your data collected will be discarded. Should 1 member of the family withdraw from the research midway, other members of the family would automatically be excluded. Data of the family unit will be discarded.

However, if you request to withdraw after the code key/personal data have been discarded, we will not be able to discard your data as we will not be able to identify which dataset belongs to whom.

### 13. Whom should I call if I have any questions or problems?

Please contact the Principal Investigator, Ms. Jamie Ong at <a href="mailto:psyoj@nus.edu.sg">psyoj@nus.edu.sg</a> for all research-related matters and in the event of research-related injuries.

For an independent opinion specifically regarding the rights and welfare of research participants, you may contact a staff member of the National University of Singapore Institutional Review Board at telephone (+65) 6516 1234 [Mondays to Thursdays from 8.30am to 6pm, and Fridays from 8.30am to 5.30pm, except public holidays] or email at irb@nus.edu.sg.





# **Parent Consent Form**

### **Protocol title:**

Exploring the Role of Parental Emotion Regulation and Outcomes of Parental Emotional Coaching on Child and Adolescent Psychosocial Outcomes

## Principal Investigator with the contact number and organization:

Principal Investigator: Ong Jiehan Jamie Organization: National University of Singapore

Email: psyoj@nus.edu.sg

My child/ward and I hereby acknowledge that:

- 1. We have agreed to take part in the above research.
- 2. We have received a copy of this information sheet that explains the use of our *data* in this research. We understand its contents and agree to donate our *data* for the use of this research.
- 3. We can withdraw from the research at any point of time by informing the Principal Investigator and all our data will be discarded. However, our data may not be able to be discard if it is no longer individually identifiable.
- 4. We will not have any financial benefits that result from the commercial development of this research.

5. We understand that our responses on the respective questionnaire sets would be kept

strictly confidential and not revealed to other members of our family.
 Yes, I am interested in attending the parent workshop (which includes 2 Zoom/phone consultation with a psychologist).
 No, I do not want to attend the parent workshop.

| Name and Signature of Participant | Relationship to Adolescent: □ Father □ Mother |
|---|---|
| Email & Contact Number | |
| Name of Child | Date |
| Name and Signature of Consent Taker | |





# Child Consent Form (for 13 years old and above)

### **Protocol title:**

Exploring the Role of Parental Emotion Regulation and Outcomes of Parental Emotional Coaching on Child and Adolescent Psychosocial Outcomes

# Principal Investigator with the contact number and organization:

Principal Investigator: Ong Jiehan Jamie Organization: National University of Singapore

Email: psyoj@nus.edu.sg

## I hereby acknowledge that:

- 1. I agree to participate in this research study.
- 2. I have read the above Information Sheet, which explains the collection and use of my information in this research.
- 3. I understand what I need to do in this research.
- 4. I know that I can withdraw from this research at any time without giving any reason by informing the investigators, and my responses will be discarded.
- 5. I understand that, unless I've given permission, my responses on the respective questionnaire sets would be kept strictly confidential and not revealed to other members of my family.

| | Yes, I agree to participate in the study. |
|------|-------------------------------------------|
| Name | of Participant |
| Name | and Signature of Consent Taker |
| Date | |